CLINICAL TRIAL: NCT04424433
Title: Myocardial Strain Analysis in Patients With Coronary Artery Disease at Hyperoxia and Normoxaemia Prior to Coronary Artery Bypass Graft Surgery - a Randomized Crossover Study
Brief Title: Myocardial Strain Analysis in Anaesthetized Coronary Artery Disease Patients During Hyperoxia and Normoxaemia
Acronym: Strecho-O₂
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-00145; SNCTP000003911 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease; Anesthesia
Keywords: Coronary artery disease; Transesophageal Echocardiography (TEE); Hyperoxia; Strain; Myocardial Deformation; Anaesthesia; CABG; Normoxaemia
MeSH Terms: conditions — Coronary Artery Disease; Hyperoxia; Sprains and Strains | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: TEE images will be coded and analysed in batches at a later date by a blinded reader
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normoxaemia First (Other): Patients will undergo TEE imaging at normoxaemia (FiO2=0.3) first, and hyperoxia (FiO2=0.8) will be targeted second.
  Interventions: Drug: Oxygen
- Hyperoxia First (Other): Patients will undergo TEE imaging at hyperoxia (FiO2=0.8) first, and normoxaemia (FiO2=0.3) will be targeted second.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Two FIO2 settings during stable general anaesthesia resulting in normoxaemic and hyperoxic arterial oxygen partial pressures.
  Other Names: Medical gas

SUMMARY:
The purpose of this study is to investigate the impact of supraphysiologic oxygen (hyperoxia) on myocardial function in anaesthetized patients with coronary artery disease.

DETAILED DESCRIPTION:
Up to 106 patients with coronary artery disease undergoing elective coronary artery bypass graft (CABG) surgery will be recruited to undergo this single visit study. In the timeframe shortly after the induction of anaesthesia and prior to the start of surgery, myocardial strain as a marker of cardiac function will be measured by transesophageal echocardiography (TEE). Echocardiography measurements will be acquired at two different oxygen states for each patient. The fraction of inspired oxygen (FiO2) will be adjusted to reach a normoxaemic state (FiO2=0.3) and a hyperoxic state (FiO2=0.8). Patients will be randomized to which oxygen level is investigated first. Thereafter, the study intervention is completed and anaesthesia and surgery will be performed as planned by the treating team. Echocardiography images will be analyzed in a blinded manner for cardiac function and systolic and diastolic strain parameters. The results will help anaesthesiologists to better weigh risks and benefits when selecting an inspired oxygen fraction in such patients, and will help to evaluate hyperoxia as a risk factor for myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG surgery (with or without other cardiac surgery)
* Ability to give and sign informed consent
* Age >18 years.

Exclusion Criteria:

* Absolute contraindication for TEE
* Emergency surgery, including but not limited to patients with instable CAD: ST- and Non-ST-elevation myocardial infarction (STEMI, NSTEMI) and instable angina (instable AP)
* Atrial fibrillation or significant arrhythmia
* Pacemaker, CRT, left bundle branch block
* Severe-grade valvular disease
* Pericardial disease
* Previous cardiac or thoracic aortic surgery
* Previous chest radiation therapy or cardiotoxic or bleomycin chemotherapy
* Severe pulmonary hypertension, cor-pulmonale, or right ventricular dysfunction, i.e., where high FIO2 might reduce pulmonary vascular resistance and right ventricular afterload
* Patients where study explanation and informed consent cannot been performed/obtained at the latest on the day before scheduled surgery
* Females of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Difference in myocardial peak strain between oxygen levels | Through study completion, within 1hour post-induction
  Percent (%), a measure of systolic function (shortening and thickening) of the myocardium

SECONDARY OUTCOMES:
Difference in myocardial time to peak strain between oxygen levels | Through study completion, within 1hour post-induction
  Milliseconds (ms)
Difference in myocardial strain rate between oxygen levels | Through study completion, within 1hour post-induction
  Change in strain over time (/second)
Difference in myocardial strain rate ratio between oxygen levels | Through study completion, within 1hour post-induction
  Change in E/A ratio
Difference in myocardial displacement between oxygen levels | Through study completion, within 1hour post-induction
  Millimeters (mm)
Difference in myocardial time to peak displacement between oxygen levels | Through study completion, within 1hour post-induction
  Milliseconds (ms)
Difference in myocardial velocities between oxygen levels | Through study completion, within 1hour post-induction
  Change in displacement over time (millimeters/second)
Difference in myocardial velocity ratio between oxygen levels | Through study completion, within 1hour post-induction
  Change in E/A ratio
Difference in peak twist | Through study completion, within 1hour post-induction
  Degrees (°)
Difference in peak torsion | Through study completion, within 1hour post-induction
  Degrees/centimeter (°/cm)
Difference in ejection fraction (EF) | Through study completion, within 1hour post-induction
  Percent (%)
Difference in chamber volumes | Through study completion, within 1hour post-induction
  Millilitres (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik P Guensch, MD, Principal Investigator — Bern University Hospital, Inselspital
Locations (1):
- Bern University Hospital, Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Guensch DP, Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, Erdoes G, Grani C, von Tengg-Kobligk H, Raber L, Eberle B. Effect of Hyperoxia on Myocardial Oxygenation and Function in Patients With Stable Multivessel Coronary Artery Disease. J Am Heart Assoc. 2020 Mar 3;9(5):e014739. doi: 10.1161/JAHA.119.014739. Epub 2020 Feb 22. PMID 32089047
- [Background] Guensch DP, Fischer K, Shie N, Lebel J, Friedrich MG. Hyperoxia Exacerbates Myocardial Ischemia in the Presence of Acute Coronary Artery Stenosis in Swine. Circ Cardiovasc Interv. 2015 Oct;8(10):e002928. doi: 10.1161/CIRCINTERVENTIONS.115.002928. PMID 26405156
- [Background] Guensch DP, Friess JO, Eberle B, Erdoes G. Hyperoxia-a Wolf in Sheep's Clothing? J Cardiothorac Vasc Anesth. 2019 May;33(5):1179-1180. doi: 10.1053/j.jvca.2018.12.024. Epub 2018 Dec 27. No abstract available. PMID 30685156
- [Background] de Jonge S, Egger M, Latif A, Loke YK, Berenholtz S, Boermeester M, Allegranzi B, Solomkin J. Effectiveness of 80% vs 30-35% fraction of inspired oxygen in patients undergoing surgery: an updated systematic review and meta-analysis. Br J Anaesth. 2019 Mar;122(3):325-334. doi: 10.1016/j.bja.2018.11.024. Epub 2019 Jan 6. PMID 30770050
- [Background] Morkane CM, McKenna H, Cumpstey AF, Oldman AH, Grocott MPW, Martin DS; Pan London Perioperative Audit and Research Network (PLAN); South Coast Perioperative Audit and Research Collaboration (SPARC). Intraoperative oxygenation in adult patients undergoing surgery (iOPS): a retrospective observational study across 29 UK hospitals. Perioper Med (Lond). 2018 Jul 24;7:17. doi: 10.1186/s13741-018-0098-3. eCollection 2018. PMID 30062007
- [Derived] Friess JO, Mikasi J, Baumann R, Ranjan R, Fischer K, Levis A, Terbeck S, Hirschi T, Gerber D, Erdoes G, Schoenhoff FS, Carrel TP, Madhkour R, Eberle B, Guensch DP. Hyperoxia-induced deterioration of diastolic function in anaesthetised patients with coronary artery disease - Randomised crossover trial. BJA Open. 2023 Apr 27;6:100135. doi: 10.1016/j.bjao.2023.100135. eCollection 2023 Jun. PMID 37588173